CLINICAL TRIAL: NCT06487936
Title: A Multi-Center, Real World Prospective/Retrospective Registry to Evaluate Patient Satisfaction With the TransLoc 3D SI Joint Fusion System
Brief Title: Real-World Registry Study on Patient Satisfaction With TransLoc 3D SI Joint Fusion
Acronym: RELIEF
Status: Recruiting | Type: Observational
Sponsor: CornerLoc (Industry)
Responsible Party: Sponsor
Other Study IDs: RELIEF-02-24
Record Dates: First submitted 2024-06-24; First posted 2024-07-05 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Sacroiliac Joint Dysfunction; Sacroiliac; Fusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Implanted TransLoc 3D SIJ Fusion Patients: Patients who were diagnosed with sacroiliitis and were treated with the TransLoc 3D System ≥ 1 year ≤ 18 months at the time of consent.
  Interventions: Device: TransLoc 3D SI Joint Fusion System

INTERVENTIONS:
Device: TransLoc 3D SI Joint Fusion System — Satisfaction survey will be administered to collect real world evidence on patients that previously received the TransLoc 3D System commercially.

SUMMARY:
This is a multi-center, consecutive enrollment registry study to evaluate patient satisfaction post SI Fusion with the TransLoc 3D SI Fusion System.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 year or older
* Confirmed Implant of the Transloc 3D Fusion System
* Did not have Transloc device removed or another manufacturer device implanted post Transloc
* Does not have other manufacturer's titanium or metal implant
* Patient may be included with prior allograft implant
* Willing to participate and give written consent
* Must have or planned CT post ≥1 year per standard of care

Exclusion Criteria:

* Patient is younger than 18 years
* Patient is unable to sign the Informed Consent
* Implant of other manufacturer's titanium or alternative metal implant
* Revision with another manufacturer's implant
* Fracture or unresolved trauma of implant side after implantation of TransLoc
* Patient unwilling to participate in Patient Satisfaction Survey
* Patient has not returned for Standard of Care follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have already received the TransLoc 3D System > 1 year postoperatively < 18 months, at the time of consent.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction Survey | Prospective 12 to 18 months post surgery
  Patient satisfaction survey administered greater than 1 year post-op: satisfaction, functional improvement, and disability as it relates to their SI joint

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) of pain | Baseline up to 1 year post surgery
  Retrospective analysis of VAS pre and post surgery, if available
Oswestry Disability Index (ODI) | Baseline up to 1 year post surgery
  Retrospective analysis of ODI pre and post surgery, if available
SAEs | Time of surgery up to 90 days post surgery
  Retrospective capture of Serious Adverse Events (SAEs) from the time of SI Fusion up to 90 days post operatively that required re-operation or in-patient hospitalization.
CT Scan Second Read (Radiological Overread) | 12 to 18 months post fusion surgery
  CT scan for placement and fusion

CONTACTS AND LOCATIONS:
Overall Officials: Lee James, DO, Principal Investigator — Advanced Orthopedic Center
Locations (1):
- Advanced Orthopedic Center, Port Charlotte, Florida, United States

IPD SHARING:
Plan to Share IPD: No